CLINICAL TRIAL: NCT04082351
Title: Evaluation of Using a Nanotechnology Structured Water Magnalife® to Achieve Controlled Blood Glucose Level in Type 2 Diabetic Patients.
Brief Title: Using Nanotechnology Structured Water to Control Blood Glucose in Type 2 Diabetic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ALI KAMAL M. SAMI (Other)
Responsible Party: Sponsor-Investigator, ALI KAMAL M. SAMI, doctor, lecturer, University of Sulaimani
Organization: University of Sulaimani (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USulaimani
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Type2 Diabetes
Keywords: Nanotechnology water; HbA1c; Type 2 Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drinking Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnalife (Active Comparator): the group of patients receiving the nanotechnology structured water
  Interventions: Dietary Supplement: Nanotechnology structured water ( Magnalife)
- Ordinary water (Placebo Comparator): the group of patients receiving ordinary water
  Interventions: Dietary Supplement: ordinary water

INTERVENTIONS:
Dietary Supplement: Nanotechnology structured water ( Magnalife) — Nanotechnology structured water ( Magnalife), is given as dietary supplement to the patients to drink it according to their weight .
  Other Names: Magnalife
  Arms: Magnalife
Dietary Supplement: ordinary water — Ordinary bottled water
  Other Names: Bottled drinking water
  Arms: Ordinary water

SUMMARY:
Type 2 DM is due to insulin resistance or low insulin secretion or sometimes a combination of both. Nanotechnology structured water is a type of water that is produced using energy field modulators to change the biological, chemical, and physical properties of water molecules and improve the bioavailability of this nano-water. Objective: To find out the effect of drinking nanotechnology structured water (Magnalife®) on the blood glucose levels in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a blind randomized control trial, according to CONSORT guidelines for randomization, "Participants were randomly assigned following simple randomization procedures (computerized random numbers) to 1 of 2 treatment groups.", that included 387 patients with Type 2 diabetes mellitus in Diabetes Care Center, Sulaymaniyah, Kurdistan region from July 2016 till February 2018. A total of 387 patients with type 2 diabetes who were patients in this center and agreed to participate in this clinical trial were included in this study.

In group A, patients were given nanotechnology structured water Magnalife® and in group B they were given ordinary bottled drinking water as a control . The bottles were unlabeled so that the patients did not know which water they were drinking. Then they were asked to eat their usual food and to drink their usual drinks, also they could drink water ad libitum after drinking the daily doses, and to have the same physical activities that they used to do in their usual daily life. They were instructed to take their medications as usual, and were told to come to test their blood sugar level at the end of the third month to get the HbA1c tested at the end of the three months of drinking the water.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients

Exclusion Criteria:

* Malignancy
* Steroids
* Immunotherapy
* Chemotherapy
* Radiotherapy
* Chronic infections
* Drugs that antagonize or synergies insulin effects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2016-07-03 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
HbA1c | three months
  measurement of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Ali K M.Sami, Ph.D., Principal Investigator — College of Medicine, University of Sulaimani

IPD SHARING:
Plan to Share IPD: Yes
The plan may include the levels of HbA1c, the medications used by the patients, the duration of their DM. But no personal data of the patients can be shared according to the agreement with patients under study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six months from the time it is public until one year after the date of being public.
Access Criteria: To obtain the IPD, an email should be sent to the investigator to ask for IPD and then get access to the plan.

REFERENCES:
- [Result] Sami AKM, Amin KH, Kurmanji MT. The Novel Use of Nanotechnology Structured Water Magnalife to Control Blood Glucose Level in Type 2 Diabetic Patients. Diabetes. 2018;67(Supplement 1):1155.